CLINICAL TRIAL: NCT03061617
Title: Comparison of Pressure-controlled Ventilation With Volume-controlled Ventilation During One-lung Ventilation
Brief Title: Comparison of Different Ventilation Mode During One-lung Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, JingCang, Professor, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: B2012-064
Record Dates: First submitted 2017-02-06; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Thoracic Surgery; One Lung Ventilation; Ventilator-Induced Lung Injury
MeSH Terms: conditions — Ventilator-Induced Lung Injury

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- volume controlled ventilation (VCV) (Other): VCV mode, tide volume 6ml/kg, f 12-14, set fixed tide volume for each breath
  Interventions: Other: VCV mode
- pressure controlled ventilation (PCV) (Experimental): PCV mode, pressure is adjusted to achieve tide volume 6ml/kg, f 12-14
  Interventions: Other: PCV mode

INTERVENTIONS:
Other: VCV mode — set fixed 6ml/kg tide volume
  Arms: volume controlled ventilation (VCV)
Other: PCV mode — adjust pressure to achieve tide volume of 6ml/kg
  Arms: pressure controlled ventilation (PCV)

SUMMARY:
It is controversial as to which ventilation mode is better in one-lung ventilation(OLV), volume controlled ventilation(VCV) or pressure controlled ventilation(PCV). This study was designed to figure out if there was any difference between these two modes on oxygenation and postoperative complications under the condition of protective ventilation(PV).

DETAILED DESCRIPTION:
This is a single center, single blinded prospective study on two different ventilation mode during one lung ventilation for patients under video assistant thoracoscopy(VATS) lobectomy. After institutional approval and written informed consent were obtained, 60 patients with primary lung cancer under VATS lobectomy in Zhongshan Hospital Fudan University were enrolled and randomized into two groups:VCV group(group V) or PCV group(group P).

Inclusion criteria were age between 18-75 years , ASA I-II, lateral decubitus position with at least 1h OLV and preoperative FEV1>50% predicted. Preoperative exclusion criteria were previous lobectomy , COPD , asthma, uncompensated cardiac disease or contraindications for epidural catheter. Intraoperative exclusion criteria were SpO2 under 90% after intratracheal suction, reconfirmation the position of double lumen tracheal tube(DLT) and recruitment maneuver of dependant lungs.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II, lateral decubitus position with at least 1h OLV and preoperative FEV1>50% predicted

Exclusion Criteria:

* Preoperative exclusion criteria were previous lobectomy , COPD , asthma, uncompensated cardiac disease or contraindications for epidural catheter. Intraoperative exclusion criteria were SpO2 under 90% after intratracheal suction, reconfirmation the position of double lumen tracheal tube(DLT) and recruitment maneuver of dependant lungs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-07; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Airway pressure Ppeak | during procedure
  Airway pressure Ppeak in cmH2O.
Airway pressure Pplat | during procedure
  Airway pressure Pplat in cmH2O.
oxygenation index | during procedure
  Oxygenation index is calculated by PaO2/FiO2. PaO2 is measured by blood-gas analysis in mmHg. FiO2 is measured by gas monitor.
oxygenation index | surgery
  Oxygenation index is calculated by PaO2/FiO2. PaO2 is measured by blood-gas analysis in mmHg. FiO2 is calculated by [21+4×oxygen flow(L/min)]×100%.

SECONDARY OUTCOMES:
postoperative complications | within 30 days after surgery
  including air leak, pneumonia, bronchopleural fistula, respiratory failure, ARDS, reintubation, tracheostomy, pulmonary embolism, arrhythmia requiring treatment, myocardial infarction, renal dysfunction, central neurologic event, sepsis, unexpected return to operating room, unexpected ICU admission and mortality within 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Song SY, Jung JY, Cho MS, Kim JH, Ryu TH, Kim BI. Volume-controlled versus pressure-controlled ventilation-volume guaranteed mode during one-lung ventilation. Korean J Anesthesiol. 2014 Oct;67(4):258-63. doi: 10.4097/kjae.2014.67.4.258. Epub 2014 Oct 27. PMID 25368784
- [Background] Lin F, Pan L, Qian W, Ge W, Dai H, Liang Y. Comparison of three ventilatory modes during one-lung ventilation in elderly patients. Int J Clin Exp Med. 2015 Jun 15;8(6):9955-60. eCollection 2015. PMID 26309682